CLINICAL TRIAL: NCT03750903
Title: Effects of Aging on Cortical Excitability During Motor Learning
Brief Title: Effect of Aging on Cortical Excitability and Motor Learning
Acronym: ACE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: E2619-R
Record Dates: First submitted 2018-11-20; First posted 2018-11-23 (Actual); Results first posted 2025-04-03 (Actual); Last update posted 2025-04-03 (Actual); Status verified 2025-04

CONDITIONS: Aging
Keywords: aging
MeSH Terms: interventions — Exercise

STUDY DESIGN:
Intervention Model Description: Two group parallel design
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Aerobic Exercise (Experimental): Participants will engage in an aerobic exercise program meeting thrice weekly for a period of 12 weeks.
  Interventions: Behavioral: Aerobic Exercise
- Stretching and Balance Training (Active Comparator): Participants will engage in a balance and stretching comparator condition meeting thrice weekly for 12 weeks.
  Interventions: Behavioral: Stretching and Balance Training

INTERVENTIONS:
Behavioral: Aerobic Exercise — Participants will engage in an aerobic exercise program meeting thrice weekly for a period of 12 weeks.
  Other Names: AE; Exercise
  Arms: Aerobic Exercise
Behavioral: Stretching and Balance Training — Participants will engage in a balance and stretching comparator condition meeting thrice weekly for 12 weeks.
  Other Names: BAL; Balance
  Arms: Stretching and Balance Training

SUMMARY:
The objective of the current proposal is to identify 1) how aging-related changes in GABAergic cortical inhibition affect motor performance, and 2) how aerobic exercise may improve inhibitory function and facilitate motor learning.

DETAILED DESCRIPTION:
The current proposal seeks quantify neural inhibition using magnetic resonance spectroscopy (MRS) and transcranial magnetic stimulation (TMS) in older Veterans to identify how each measures contributes to aging-related changes in motor performance. Currently, over 56% (11.8 million) of Veterans are over age 60. Recent research has shown that aging is associated with decreased cortical inhibition and impaired hand motor function. However, this loss of inhibition is not an inescapable consequence of aging. The investigators' previous work that healthy older adults who engage in regular physical activity show increased cortical inhibition and improved dexterity as compared to their sedentary age cohort. This indicates that aerobic training may reverse aging related changes in cortical inhibition and alteration of tonic levels of cortical excitability can have a powerful impact on motor performance in the aging brain. In the current proposal, the investigators will enroll older adults to assess how different measurements (TMS and MRS) of the dominant inhibitory neurotransmitter in the brain - GABA differ in relation to motor control. During the MRS scan, participants will perform a motor learning task to assess change in GABA level throughout the acquisition session. These data will be compared with measures of cortical inhibition using TMS to quantify neurotransmitter receptor activity with respect to aging-related changes in motor performance. The investigators will also be comparing the effects of an aerobic exercise intervention as compared to a contact matched stretching control. The investigators believe this project is the first inquiry of its kind and will have an important impact in the understanding of aging-related neurophysiological changes in the brain and how it can remediate associated behavioral declines.

ELIGIBILITY:
Inclusion Criteria:

* living persons aged 50-85

Exclusion Criteria:

* unmanaged diabetes
* participants completing vigorous exercise per week
* participants whose profession requires vigorous physical labor
* contraindication to magnetic resonance imaging

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2019-03-04 (Actual); Primary Completion 2023-09-30 (Actual); Study Completion 2024-09-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joe R. Nocera, PhD, Principal Investigator — Atlanta VA Medical and Rehab Center, Decatur, GA
Locations (1):
- Atlanta VA Medical and Rehab Center, Decatur, GA, Decatur, Washington, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Aerobic Exercise | Stretching and Balance Training
Started | 12 | 18
Completed | 10 | 10
Not Completed | 2 | 8

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Aerobic Exercise | Stretching and Balance Training | Total
Number analyzed (Participants) | 12 | 18 | 30
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 12 | 18 | 30
Age, Continuous [Mean (Full Range); unit: years] | 69.88 [66 to 76] | 71.24 [65 to 80] | 70.02 [65 to 80]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 10 | 16
  Male | 6 | 8 | 14
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 5 | 10 | 15
  White | 6 | 7 | 13
  More than one race | 0 | 1 | 1
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 12 | 18 | 30

OUTCOME MEASURES:

1. Primary Outcome: Magnetic Resonance Spectroscopy
Description: Measuring changes in dynamic magnetic resonance spectroscopy of primary motor cortex during motor learning.
Time Frame: Baseline and12 weeks
Population: 4 participants in the Aerobic exercise group and 10 participants in the Stretching and Balance Training group did not complete the 12 week follow up assessment
Measure: Mean (Standard Deviation); unit: ppm
Arm/Group | Aerobic Exercise | Stretching and Balance Training
Number analyzed (Participants) | 8 | 8
ppm | 0.41 (0.69) | -0.29 (0.66)
Statistical Analysis 1: Comparison: Aerobic Exercise vs Stretching and Balance Training; Test type: Other; p = 0.05, ANOVA

ADVERSE EVENTS:
Time Frame: 14 weeks from baseline assessment through 12-week intervention to follow up assessment.
Arm/Group | Aerobic Exercise | Stretching and Balance Training
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/18
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/18
Other Adverse Events (participants affected / at risk) | 0/12 | 0/18

LIMITATIONS AND CAVEATS:
COVID-19 impacted the in person exercise interventions

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-08-30): https://cdn.clinicaltrials.gov/large-docs/03/NCT03750903/Prot_SAP_000.pdf
  • Informed Consent Form (2021-11-26): https://cdn.clinicaltrials.gov/large-docs/03/NCT03750903/ICF_001.pdf